CLINICAL TRIAL: NCT07251738
Title: Understanding the Lived Experience and Bereavement of Caregivers of People With Alzheimer's Disease
Acronym: ALCARE
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Sara Garcia Bravo, PhD Physiotherapist, Universidad Rey Juan Carlos
Other Study IDs: 041220246522024
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease (AD); Occupational Therapy; Family Caregivers
Keywords: Alzheimer's disease; Occupational Therapy; occupational balance
MeSH Terms: conditions — Alzheimer Disease | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: relatives of people diagnosed with AD by a neurologist or geriatrician, who have suffered the loss of a relative with AD; who have lived with and/or cared for the person with AD until the end of their life
  Interventions: Other: Assessment of occupational balance, role performance, caregiving burden, and quality of life among carers or family members of individuals with Alzheimer's disease (AD).
- Group 2: relatives of people diagnosed with AD by a neurologist or geriatrician; who lived with and/or cared for the person with AD; who attended the Day Centre
  Interventions: Other: Assessment of occupational balance, role performance, caregiving burden, and quality of life among carers or family members of individuals with Alzheimer's disease (AD).
- Group 3: relatives of people diagnosed with AD by a neurologist or geriatrician; who had their relative institutionalised in the Residence
  Interventions: Other: Assessment of occupational balance, role performance, caregiving burden, and quality of life among carers or family members of individuals with Alzheimer's disease (AD).

INTERVENTIONS:
Other: Assessment of occupational balance, role performance, caregiving burden, and quality of life among carers or family members of individuals with Alzheimer's disease (AD). — Assessment of occupational balance, role performance, caregiving burden, and quality of life among carers or family members of individuals with Alzheimer's disease (AD).

SUMMARY:
The main objective of this study is to explore the lived experience of caregivers and family members of people with Alzheimer's disease (AD), from the beginning of caregiving through the bereavement process following the patient's death. Using a mixed-methods design, qualitative data will be collected through in-depth interviews and combined with quantitative data obtained from standardized scales. The results will aim to determine whether prolonged caregiving significantly affects the caregiver's or family member's personal, emotional, and occupational well-being, as well as whether it leads to a reorganization of activities of daily living (ADL), an increased perception of burden, and/or a decreased quality of life. The study will also examine the presence of positive adaptation experiences.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for Group 1: relatives of people diagnosed with AD by a neurologist or geriatrician, who have suffered the loss of a relative with AD; who have lived with and/or cared for the person with AD until the end of their life; who agree to participate voluntarily in the project and who have signed the informed consent form.
* Inclusion criteria for Group 2: relatives of people diagnosed with AD by a neurologist or geriatrician; who live with and/or care for the person with AD; who attend the Day Centre and who agree to participate voluntarily in the project and have signed the informed consent form.
* Inclusion criteria for Group 3: relatives of people diagnosed with AD by a neurologist or geriatrician; who have their relative institutionalised in a nursing home and who agree to participate voluntarily in the project and have signed the informed consent form.

Exclusion Criteria:

* Those who have not lived with or cared for relatives with AD and who do not agree to participate in the study will be excluded from the project.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: relatives of individuals diagnosed with AD by a neurologist or geriatrician
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Zarit Burden Interview, ZBI | baseline
  is a tool designed to assess the level of perceived burden experienced by informal carers of dependent persons. It consists of 22 items that explore emotional, social and physical aspects related to caregiving, allowing the impact of the carer role on their quality of life to be identified. Each item is scored on a Likert scale, with higher scores indicating greater burden.
Role Checklist | baseline
  It is an instrument based on the Human Occupation Model (HOM) designed to assess the occupational roles that a person performs throughout their life. It allows for the identification of current, past, and future roles, as well as the subjective value assigned to each one. This instrument is useful for understanding how occupational roles contribute to a sense of identity, the organisation of daily life and overall well-being, facilitating the planning of client-centred interventions.
Short Form-36 Health Survey | baseline
  It is a widely used tool for measuring health-related quality of life. It assesses eight dimensions: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. It is a generic instrument, applicable to diverse populations and useful in both research and practice, providing a broad profile of people's health status.
Occupational Balance Questionnaire | baseline
  It is an assessment tool designed to measure occupational balance, understood as people's perception of the appropriate distribution of their time and energy in meaningful activities. This questionnaire explores aspects related to satisfaction and management of daily occupations, considering both the quantity and quality of the activities performed. It has proven useful in clinical and research contexts to identify occupational imbalances that can affect health and well-being. The original version was developed in Sweden and has been adapted to various languages and cultures, maintaining its validity and reliability.

IPD SHARING:
Plan to Share IPD: No